CLINICAL TRIAL: NCT04799743
Title: A Pilot Randomized Controlled Clinical Study of Resveratrol for Discharged COVID 19 Patients in Order to Evaluate Its Therapeutic Effects Against Fibrosis
Brief Title: The Anti-fibrotic Therapeutic Effects of Resveratrol for Discharged COVID-19 Patients
Acronym: HKCOVID19Res
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hong Kong Baptist University (Other)
Collaborators: Hospital Authority, Hong Kong (Other Government)
Responsible Party: Principal Investigator, Zhong Lidan, Assistant Professor, Hong Kong Baptist University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HKCOVID19Resveratrol
Record Dates: First submitted 2021-03-10; First posted 2021-03-16 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Covid-19
Keywords: rehabilitation; Chinese medicine; randomized controlled trial
MeSH Terms: conditions — COVID-19 | interventions — Resveratrol; Drug Evaluation

STUDY DESIGN:
Intervention Model Description: Randomized, Double-Blind, Placebo-Controlled Parallel Group Clinical Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The participants will be randomly assigned to resveratrol group and placebo group with 1:1 ratio. Block randomization with block size of 6 will be carried out in 1:1 ratio according to the sequence generated with Random Allocation Software (Version 2.0.0), Isfahan, Iran. Treatments will be assigned according to the codes which are kept in opaque sealed envelopes with consecutive randomization numbers. Treatment assignments will not be revealed and blinded to patients and PI (outcome assessor) until the whole study is completed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resveratrol group (Experimental): Resveratrol group (treatment group) will be instructed to consume with capsules (1.0 g, orally once a day) for six months.
  Interventions: Drug: Resveratrol
- Placebo group (Placebo Comparator): Placebo group (control group) will be instructed to orally take placebo (edible paraffin, 1.0) once a day.
  Interventions: Drug: Placebo capsules

INTERVENTIONS:
Drug: Resveratrol — Resveratrol has been used as a food supplement. Its antiviral properties have been well studied including its inhibitory effect against the coronavirus MERS-CoV. Our previous in vitro and in vivo studies found that the compound had other health benefits such as anti-fibrotic effect.The anti-fibrotic effect will add an extra benefit for resveratrol to fight against COVID-19 as lungs are the most affected organs by the coronavirus, which may result in prolonged fibrotic damage of the lungs even when a patient is recovered from the COVID-19 disease.
  Other Names: Resveratrol Capsule
  Arms: Resveratrol group
Drug: Placebo capsules — The placebo consist of mainly starch and microcrystalline cellulose, the usage and dosage are the same as the investigational drug.
  Other Names: Study drug
  Arms: Placebo group

SUMMARY:
A randomized controlled trial (RCT) will be conducted to evaluate the anti-fibrotic therapeutic effects of resveratrol on the clinical symptoms in discharged COVID-19 patients.

DETAILED DESCRIPTION:
The proposed study will be a randomized controlled trial (RCT) to evaluate the anti-fibrotic therapeutic effects of resveratrol on the clinical symptoms in discharged COVID-19 patients. The target population will be post-discharge patients recovering from COVID-19. Eligible participants will be recruited from the ongoing special Chinese Medicine program for discharged patients collaborated with Hong Kong Hospital Authority. Thirty (30) participants will be randomly assigned to resveratrol group and placebo group with 1:1 ratio. The participants will receive six months of treatment (1 g, orally and once daily) and three months of follow-up. The total duration of the clinical study is 9 months. The study protocol will be submitted to the Ethics Committee for review and approval. Participants will be enrolled and signed written informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be the patients aged 18-65 years old who have been previously diagnosed to be infected with COVID-19 and discharged from local hospitals after treatment with western medicines, and with negative results from COVID-19 virus detection. The subjects will be evaluated for potential pulmonary fibrosis and those who present with the condition resulting from COVID-19 infection will be included.

Exclusion Criteria:

* Participants will be excluded if they have one or more of the followings: 1) inability to communicate (e.g. cognitive impairment); 2) history of Chinese medicine allergies; 3) incompetent in giving consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
The handheld basic spirometry | 9 months
  Lung function will be assessed by the handheld basic spirometry (forced expiratory volume, FEV and forced vital capacity, FVC). FEV is the parameter to measure how much air the participants can force from their lungs in one second. Lower FEV-1 readings indicate more significant obstruction. FVC is the largest amount of air that the participants can forcefully exhale after breathing in as deeply as they can. A lower than normal FVC reading indicates restricted breathing. The participants will be trained to check these measurements at home and record the data in the patient diary.
PRO scores | 9 months
  All the symptoms will be measured by PRO scores according to the clinical symptoms of COVID-19 rehabilitation patients. The scores will be ranged from 0-4: "0" indicates none; "1" indicates mild; "2" indicates moderate; "3" indicates moderately severe; and '4" indicates severe.
Borg Category-Ratio 0-10 Scale | 9 months
  We will also use Borg Category-Ratio 0-10 Scale (Borg CR10 Scale) to measure dyspnea as recommended by the American College of Sports Medicine (ACSM) guidelines for patients with pulmonary diseases (Asha et al., 2012). The Borg Category Ratio 10 (CR10) Scale® (Borg Dyspnea Scale), will be used to rate the patients' dyspnea and overall fatigue level.
  Scale:
  0=Rest; 0.5=Really Really Easy; 1=Really Easy; 2=Easy; 3=Moderate; 4=Sort of Hard; 5,6=Hard; 7,8,9=Really Hard; 10=Maximal

SECONDARY OUTCOMES:
Lung Function Questionnaire with 6-min walk-test | 9 months
  Lung Function Questionnaire is a simple, brief, self-administered instrument to identify patients appropriate for lung function evaluation by 5 items about the breathing problems and/or frequent cough. It was validated in Chinese and widely used in primary care (Hanania et al., 2010).
the World Health Organization Quality of Life Brief Assessment [WHOQOL-BREF (HK)] | 9 months
  WHOQOL-BREF (HK) (Leung, K F., et al., 2005) was validated in Hong Kong and widely use in academia and clinicians since 1997. This is a 5-point Likert scale with a total of 28 Questions to identify the perceived QOL of the participants. There are four domains namely Physical Health, Psychological, Social and Environment domains with a maximum of 100.
Body constitution questionnaires | 9 months
  In 2009, the classification of body constitutions into nine specific types has been recognized by China Association of Chinese Medicine as the standard of body constitution (China Association of Chinese Medicine, 2009). Our research team also validated this questionnaire in Cantonese. The related version of questionnaire will be applied in this study. It is a self-rating scale with good reliability and validity. It contains nine subscales: gentleness, qi-deficiency, yang-deficiency, yin-deficiency, phlegm-dampness, dampness-heat, blood-stasis, qi-depression, and special diathesis. Score of each subscale is standardized from 0 to 100. Gentleness type is a balanced one with higher score indicating a better constitution status, while the other eight types are pathological types with higher score indicating worse constitution status.

CONTACTS AND LOCATIONS:
Overall Officials: Bian Zhaoxiang, MD.,PH.D, Study Director — Hong Kong Chinese Medicine Clinical Study Centre
Locations (1):
- Linda Zhong, Kowloon Tong, Kowloon, Hong Kong